CLINICAL TRIAL: NCT05647928
Title: Retinal Redetachment After Silicone Oil Removal : a Risk Factor Analysis
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Professeur Jean-Baptiste CONART, MD PhD, Central Hospital, Nancy, France
Other Study IDs: 2022PI084
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Retinal Redetachment After Silicone Oil Removal
Keywords: rhegmatogenous retinal detachment; silicone oil; proliferative vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retinal redetachment after silicone oil removal
  Interventions: Other: no intervention
- NO retinal redetachment after silicone oil removal
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To report the rate of retinal redetachment after silicone oil removal (SOR) following rhegmatogenous retinal detachment (RRD) surgery and to determine potential risk factors

ELIGIBILITY:
Inclusion Criteria:

* patients with successfully repaired rhegmatogenous retinal detachment and subsequent silicone oil removal
* minimum follow-up period of 6 months after silicone oil removal

Exclusion Criteria:

* Silicone oil tamponade for indications other than rhegmatogenous retinal detachment
* Retinal redetachment during silicone oil tamponade
* Prior history of silicone oil tamponade

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent pars plana vitrectomy with silicone oil tamponade at the Nancy University Hospital from January 2015 to January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
rate of retinal redetachment after silicone oil removal | a minimum period of 6 months after silicone oil removal
pre- and intraoperative risk factors of retinal redetachment after silicone oil removal | a minimum period of 6 months after silicone oil removal

SECONDARY OUTCOMES:
final retinal reattachment rate | a minimum period of 6 months after silicone oil removal
final best corrected visual acuity | a minimum period of 6 months after silicone oil removal

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy Brabois, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Gisquet C, Ndiaye NC, Dubroux C, Angioi-Duprez K, Berrod JP, Conart JB. Retinal redetachment after silicone oil removal: a risk factor analysis. BMC Ophthalmol. 2024 Aug 15;24(1):346. doi: 10.1186/s12886-024-03618-z. PMID 39148018